CLINICAL TRIAL: NCT01596595
Title: Longitudinal Surveillance Study of the 4-SITE Lead/Header System
Acronym: LSS of 4-SITE
Status: Completed | Type: Observational
Sponsor: Boston Scientific Corporation (Industry)
Responsible Party: Sponsor
Other Study IDs: LSS of 4-SITE
Record Dates: First submitted 2012-05-03; First posted 2012-05-11 (Estimated); Results first posted 2021-02-21 (Actual); Last update posted 2021-03-19 (Actual); Status verified 2021-02

CONDITIONS: Primary Prevention of Sudden Cardiac Arrest; Secondary Prevention of Sudden Cardiac Arrest
Keywords: ICD; CRT-D; Defibrillation lead

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Medically Indicated for ICD or CRT-D: Medically Indicated for ICD or CRT-D implantation per guidelines

SUMMARY:
Post-approval studies of implanted leads provide an opportunity to observe and assess patient outcomes and technology performance in a real-world setting. The goal of the study is to evaluate, document and report on the appropriate clinical performance, long-term reliability and the functional integrity of the Boston Scientific ENDOTAK RELIANCE® 4-SITE™ Lead and the pulse generator 4-SITE Header.

DETAILED DESCRIPTION:
The objective of the LSS of 4-SITE Study is to prospectively determine the chronic complication-free rate of the 4-SITE Lead/Header System in order to verify its clinical performance, long-term reliability and functional integrity. The LSS of 4-SITE Study is a non-randomized, multi-center, global clinical investigation of subjects implanted with the 4-SITE Lead/Header System. The study is designed to collect product performance information, any reportable adverse events and withdrawal data.

The primary purpose of this study is to evaluate, document and report on the appropriate clinical performance, the long-term reliability and the functional integrity of the 4-SITE Lead/Header System. This 4-SITE Lead/Header System consists of a 4-SITE ENDOTAK® RELIANCE defibrillation lead connected to a 4-SITE Header (which is the only PG component under study) of a single or dual chamber (VR and DR) implantable cardioverter defibrillator (ICD) or a cardiac resynchronization therapy ICD (CRT-D) BSC pulse generator. Additionally, system-related diagnostic information and implant data will be collected during the conduct of this study.

ELIGIBILITY:
Inclusion Criteria:

* medically indicated for ICD/CRT-D
* received/plan to receive study lead
* willing for long-term follow-up

Exclusion Criteria:

* unwilling to comply with protocol

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: From Physicians patient population
Sampling Method: Non-Probability Sample
Enrollment: 1820 (Actual)
Dates: Start 2013-04-04 (Actual); Primary Completion 2020-02-18 (Actual); Study Completion 2020-02-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Kutalek, MD, Principal Investigator — Drexel University, USA
Locations (111):
- United States (104):
  - Providence Alaska Medical Center, Anchorage, Alaska
  - Cardiovascular Consultants, LTD, Glendale, Arizona
  - Cardiovascular Associates of Mesa, Mesa, Arizona
  - Phoenix Cardiovascular Research Group, Phoenix, Arizona
  - Heart Clinic Arkansas, Little Rock, Arkansas
  - Providence St. Joseph Medical Center, Burbank, California
  - Palomar Medical Center, Escondido, California
  - California Heart Associates, Fountain Valley, California
  - Luc Sinh Nguyen, MD, FACC, Inc., Fountain Valley, California
  - Providence Holy Cross Medical Center, Los Angeles, California
  - Cardiac Device Rhythm Specialists, Los Angeles, California
  - Comprehensive Cardiovascular Medical Group, Los Angeles, California
  - Desert Regional Medical Center, Palm Springs, California
  - Truong D. Duong, MD. A Medical Corporation, Riverside, California
  - San Diego Arrhythmia Associates, San Diego, California
  - Good Samaritan Hospital - San Jose, San Jose, California
  - Santa Barbara Cottage Hospital, Santa Barbara, California
  - Little Company of Mary Hospital, Torrance, California
  - University of Colorado Hospital, Aurora, Colorado
  - South Denver Cardiology Associates, PC, Denver, Colorado
  - Danbury Hospital, Danbury, Connecticut
  - Yale University School of Medicine, New Haven, Connecticut
  - Bradenton Cardiology, Bradenton, Florida
  - Clearwater Cardiovascular Consultants, Clearwater, Florida
  - Broward General Medical Center, Fort Lauderdale, Florida
  - North Florida Regional Medical Center, Gainesville, Florida
  - First Coast Cardiovascular, Jacksonville, Florida
  - Baptist Medical Center, Jacksonville, Florida
  - Osceola Regional Medical Center, Kissimmee, Florida
  - Cardiovascular Research Center of South Florida, Miami, Florida
  - Charlotte Heart & Vascular, Port Charlotte, Florida
  - Brevard Cardiovascular Research Associates, Inc., Rockledge, Florida
  - Tallahassee Memorial Hospital, Tallahassee, Florida
  - Tampa General Hospital, Tampa, Florida
  - Phoebe Putney Memorial Hospital, Albany, Georgia
  - Northeast Georgia Heart Center, Gainesville, Georgia
  - Gwinnett Hospital System Inc., Lawrenceville, Georgia
  - Georgia Arrhythmia Consultants, Macon, Georgia
  - Atlanta Heart Associates, Stockbridge, Georgia
  - University of Chicago Hospital, Chicago, Illinois
  - Illinois Heart and Vascular at Adventist Hinsdale Hospital, Hinsdale, Illinois
  - Heartland Cardiovascular Center, Joliet, Illinois
  - Carle Foundation Hospital, Urbana, Illinois
  - Bloomington Hospital, Bloomington, Indiana
  - Parkview Memorial Hospital, Fort Wayne, Indiana
  - Mercy Hospital Medical Center, Des Moines, Iowa
  - The Iowa Clinic, PC, Des Moines, Iowa
  - Kansas City Heart Foundation, Kansas City, Kansas
  - Via-Christi Regional Medical Center, Wichita, Kansas
  - Ochsner Clinic Foundation, New Orleans, Louisiana
  - University of Maryland Medical System, Baltimore, Maryland
  - MedStar Health Research Institute, Baltimore, Maryland
  - University of Massachusetts Memorial Medical Center, Worcester, Massachusetts
  - St. Joseph Mercy Hospital, Ann Arbor, Michigan
  - Covenant Medical Center, Saginaw, Michigan
  - Munson Medical Center, Traverse City, Michigan
  - Centracare Heart and Vascular Center, Saint Cloud, Minnesota
  - University of Mississippi Medical Center, Jackson, Mississippi
  - North Mississippi Medical Center, Tupelo, Mississippi
  - Cox Health, Springfield, Missouri
  - St. Louis University Hospital, St Louis, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Billings Clinic, Billings, Montana
  - St. Patrick Hospital, Missoula, Montana
  - Nebraska Heart Institute, Lincoln, Nebraska
  - Deborah Heart and Lung Center, Browns Mills, New Jersey
  - Englewood Hospital and Medical Center, Englewood, New Jersey
  - Cardiovascular Associates of the Delaware Valley, Sewell, New Jersey
  - North Shore University Hospital, Manhasset, New York
  - Rochester General Hospital, Rochester, New York
  - SUNY-Stony Brook School of Medicine, Stony Brook, New York
  - Cardiology Group of West New York, Williamsville, New York
  - Universtity of Cincinnati, Cincinnati, Ohio
  - University Hospitals of Cleveland, Cleveland, Ohio
  - Kettering Medical Center, Kettering, Ohio
  - The Toledo Hospital, Toledo, Ohio
  - Genesis Healthcare System, Zanesville, Ohio
  - Salem Hospital, Salem, Oregon
  - The Arrhythmia Institute, Newton, Pennsylvania
  - Drexel University College of Medicine, Philadelphia, Pennsylvania
  - Cardiology Consultants of Philadelphia, Yardley, Pennsylvania
  - Southcoast Physicians Group, Providence, Rhode Island
  - Sisters of Charity Providence Hospital, Columbia, South Carolina
  - PeeDee Cardiology Associates PA, Florence, South Carolina
  - Piedmont Medical Center, Greenwood, South Carolina
  - Lexington Medical Center, Lexington, South Carolina
  - Spartanburg Regional Medical Center, Spartanburg, South Carolina
  - Rapid City Regional Hospit, Rapid City, South Dakota
  - Saint Thomas Health, Nashville, Tennessee
  - Wellmont Holston Valley Medical Center, Rogersville, Tennessee
  - SouthEast Texas Clinical Research Center, Beaumont, Texas
  - Houston Arrhythmia Associates, Houston, Texas
  - Arrhythmia Associates of South Texas, San Antonio, Texas
  - Trinity Mother Frances Health System, Tyler, Texas
  - Intermountain Medical Center, Murray, Utah
  - University of Utah Hospital and Clinics, Salt Lake City, Utah
  - Sentara Norfolk General Hospital, Norfolk, Virginia
  - Virginia Commonwealth University Health System, Richmond, Virginia
  - Virginia Mason Medical Center, Seattle, Washington
  - Charleston Area Medical Center, Charleston, West Virginia
  - Monongalia General Hospital, Morgantown, West Virginia
  - Bellin Health, Green Bay, Wisconsin
  - Meriter Hospital, Inc., Madison, Wisconsin
  - Cheyenne Regional Medical Center, Cheyenne, Wyoming
- Mount Hospital, Perth, Western Australia, Australia
- Canada (6):
  - Foothills Medical Centre, Calgary, Alberta
  - University of Alberta Hospital, Edmonton, Alberta
  - Royal Columbian Hospital, New Westminster, British Columbia
  - Hamilton General Hospital, Hamilton, Ontario
  - Fleurimont Hospital, Sherbrooke, Quebec
  - Institut universitaire de Cardiologie et de Pneumologie de Quebec, Ste Foy, Quebec

RESULTS

PARTICIPANT FLOW:
Groups:
- RELIANCE 4-SITE: There were 1820 patients who were consented for participation in the LSS of 4-SITE Study. Of the 1820 participants enrolled 1779 were implanted and followed for the study. There were 11 subjects who were attempted for implant but did not receive a study devices and 30 subjects who were determined to be intent subjects (did not undergo surgery) and were withdrawn from the study.
Period: Overall Study
Arm/Group | RELIANCE 4-SITE
Started | 1779
Completed | 814
Not Completed | 965

BASELINE CHARACTERISTICS:
Population: Baseline characteristics include enrolled subjects who were implanted (1779) or attempted for implant (11) of an ENDOTAK® RELIANCE 4-SITE lead and Boston Scientific pulse generator compatible with the RELIANCE 4-SITE family of cardiac leads. Intent subjects (30) are not included in the baseline characteristics.
Groups:
- RELIANCE 4-SITE: Baseline characteristics include enrolled subjects who were implanted (1779) or attempted for implant (11) of an ENDOTAK® RELIANCE 4-SITE lead and Boston Scientific pulse generator compatible with the RELIANCE 4-SITE family of cardiac leads. Intent subjects (30) are not included in the baseline characteristics.
Arm/Group | RELIANCE 4-SITE
Number analyzed (Participants) | 1790
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.0 (12.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 481
  Male | 1309
Race/Ethnicity, Customized [Number; unit: Participant selections] — Participants may contribute to more than one category.
  Participant selections
    Caucasian | 1345
    Black | 249
    Hispanic | 106
    Not Disclosed | 39
    Asian | 24
    American Indian or Alaska Native | 19
    Hawaiian | 2
    Other | 7
    Missing data | 8
Region of Enrollment [Number; unit: participants]
  Canada | 107
  United States | 1681
  Australia | 2

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Not Experiencing a System or Procedure Related Complication Through 5-years
Description: The 4-SITE Lead/Header System will be evaluated based on the "chronic 4-SITE Lead/Header System-related complication-free rate" for the five (5) year follow-up period after the index implantation. The primary endpoint analysis will include confirmed chronic 4-SITE Lead/Header System-related complications that result in study subject permanent loss of therapy, invasive intervention, injury or death.
Time Frame: 5 years
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Groups:
- RELIANCE 4-SITE: There were 1820 patients who were consented for participation in the LSS of 4-SITE Study. Of the 1820 participants enrolled 1779 were implanted and followed for the study. There were 11 subjects who were attempted for implant but did not receive a study devices and 30 subjects who were determined to be intent subjects (did not undergo surgery) and were withdrawn from the study. These 41 subjects are not included in the endpoint analysis. The endpoint was analyzed using intent to treat analysis.
Arm/Group | RELIANCE 4-SITE
Number analyzed (Participants) | 1779
Percentage of participants | 98.9 [98.5 to NA] — As prespecified in the study protocol the lower one-sided 95% confidence bound of the Kaplan-Meier estimate was compared to the performance goal (i.e., only the lower one-side confidence bound was necessary/utilized for hypothesis testing).

ADVERSE EVENTS:
Time Frame: Adverse event data were collected from the time of enrollment until subjects ended their participation in the study. Subjects were considered to have completed the study after 60-Months of follow-up.
Groups:
- RELIANCE 4-SITE: All-Cause Mortality and Adverse Events are reported for all enrolled subjects (N=1820).
Arm/Group | RELIANCE 4-SITE
All-Cause Mortality (participants affected / at risk) | 327/1820
Serious Adverse Events (participants affected / at risk) | 1017/1820
Other Adverse Events (participants affected / at risk) | 980/1820
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | RELIANCE 4-SITE (N=1820)
Other - PG System (Product Issues) | 2
Elevated Threshold - RV (Product Issues) | 1
Inappropriate Tachy Therapy - SVT (Product Issues) | 30
Inappropriate Tachy Therapy - Other (Product Issues) | 6
Early ERI - Premature Declaration (Product Issues) | 1
Pacemaker Mediated Tachycardia (PMT) (Product Issues) | 2
Erosion (Product Issues) | 2
Infection (> 30 days post implant) (Infections and infestations) | 8
Hematoma- Pocket (>30 days post implant) (Injury, poisoning and procedural complications) | 1
Migration (Injury, poisoning and procedural complications) | 1
Post Surgical wound discomfort/bruising/swelling (Injury, poisoning and procedural complications) | 3
Post-surgical pocket hemorrhage/bleeding/drainage (Injury, poisoning and procedural complications) | 1
Post -Surgical infection (≤ 30 days post implant) (Injury, poisoning and procedural complications) | 3
Adverse Reaction - Respiratory (Injury, poisoning and procedural complications) | 2
Chest pain (Injury, poisoning and procedural complications) | 5
Hematoma - pocket (≤ 30 days post-implant) (Injury, poisoning and procedural complications) | 8
Thromboembolic events (Injury, poisoning and procedural complications) | 4
Procedure - PG System - Other (Injury, poisoning and procedural complications) | 1
Dislodgement - Unable to Capture - RA (Product Issues) | 1
Dislodgement - Multiple signs- RA (Product Issues) | 1
Dislodgement - No reported signs - RA (Product Issues) | 4
Other Lead Related (Product Issues) | 3
Oversensing - RV (Product Issues) | 1
Unable to Capture - RV (Product Issues) | 3
Elevated Threshold - RV 2140 - Extracardiac Stimulation - RV (Product Issues) | 3
Extracardiac Stimulation - RV (Product Issues) | 1
Insulation Breach - RV (Product Issues) | 2
Myocardial Perforation post implant- RV (Product Issues) | 3
Low Out of Range Impedance - RV (Product Issues) | 1
Dislodgement - Unable to capture - RV (Product Issues) | 3
Dislodgement - Elevated threshold - RV (Product Issues) | 4
Dislodgement - Extracardiac stimulation - RV (Product Issues) | 1
Dislodgement - Multiple signs - RV (Product Issues) | 1
Dislodgement - No reported signs - RV (Product Issues) | 4
Unable to Capture - LV (Product Issues) | 1
Extracardiac Stimulation - LV (Product Issues) | 3
Conductor Coil Fracture - LV (Product Issues) | 1
Insulation Breach - LV (Product Issues) | 1
Dislodgement - Unable to Capture - LV (Product Issues) | 4
Dislodgement - Elevated threshold - LV (Product Issues) | 1
Dislodgement - Extracardiac stimulation - LV (Product Issues) | 1
Dislodgement - Multiple signs - LV (Product Issues) | 1
Dislodgement - No reported signs - LV (Product Issues) | 7
Inappropriate tachy therapy - SVT (Product Issues) | 2
Pneumothorax (Injury, poisoning and procedural complications) | 6
Hemothorax (Injury, poisoning and procedural complications) | 2
Myocardial perforation without tamponade (Injury, poisoning and procedural complications) | 1
Myocardial perforation with tamponade (Injury, poisoning and procedural complications) | 1
Pericardial Effusion (Injury, poisoning and procedural complications) | 3
Procedure - Lead - Other (Injury, poisoning and procedural complications) | 1
3rd Degree AV Block (Cardiac disorders) | 1
Sinus Bradycardia (Cardiac disorders) | 5
Pulseless Electrical Activity (PEA) (Cardiac disorders) | 13
Ventricular Fibrillation (VF) (Cardiac disorders) | 29
Ventricular Tachycardia (VT)/Monomorphic VT (Cardiac disorders) | 72
Torsades de Pointes (Cardiac disorders) | 1
Nonsustained ventricular tachycardia (NSVT) (Cardiac disorders) | 6
Atrial Fibrillation (AF) (Cardiac disorders) | 83
Atrial Flutter (Cardiac disorders) | 15
Sinus Tachycardia (Cardiac disorders) | 1
Atrial Tachycardia/Other SVT (e.g. AVRT, AVNRT, EAT) (Cardiac disorders) | 10
Premature Ventricular Contractions (PVC) (Cardiac disorders) | 2
Syncope - Heart Failure (Cardiac disorders) | 1
Dizziness - Heart Failure (Cardiac disorders) | 1
Chest Pain - Heart Failure (Cardiac disorders) | 7
Dyspnea - Heart Failure (Cardiac disorders) | 108
Peripheral edema - Heart Failure (Cardiac disorders) | 10
Pulmonary Edema - Heart Failure (Cardiac disorders) | 15
Fatigue - Heart Failure (Cardiac disorders) | 1
Renal Failure/Insufficiency - Heart Failure (Cardiac disorders) | 12
Dehydration - Heart Failure (Cardiac disorders) | 2
Gastrointestinal - Heart Failure (Cardiac disorders) | 4
Hypotension - Heart Failure (Cardiac disorders) | 4
Weight Gain - Heart Failure (Cardiac disorders) | 16
Heart Failure Symptoms - Unspecified (Cardiac disorders) | 142
Multiple Heart Failure Symptoms (Cardiac disorders) | 185
Hypertension - Heart Failure (Cardiac disorders) | 2
Heart Failure Patient Condition - Cardiovascular - OTHER (Cardiac disorders) | 6
Multi-system Failure - Heart Failure (Cardiac disorders) | 13
Hypotension/Orthostatic Hypotension (Vascular disorders) | 37
Hypertension/Hypertensive Crisis (Vascular disorders) | 11
Cardiogenic Shock (Cardiac disorders) | 20
Cardiac Arrest (Cardiac disorders) | 41
Myocardial Infarction (Vascular disorders) | 62
Peripheral Vascular Disease (Vascular disorders) | 38
Intermittent Claudication (Vascular disorders) | 2
Aortic Stenosis (Cardiac disorders) | 9
Aortic Regurgitation (Cardiac disorders) | 1
Mitral Stenosis (Cardiac disorders) | 1
Mitral Regurgitation (Cardiac disorders) | 9
Syncope (General disorders) | 37
Dizziness (General disorders) | 23
Chest Pain - Ischemic (Vascular disorders) | 19
Chest Pain - Other (General disorders) | 68
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 12
Palpitations (Cardiac disorders) | 1
Fatigue/Weakness (General disorders) | 2
Multiple Symptoms (General disorders) | 5
Patient Condition - Cardiovascular - OTHER (Cardiac disorders) | 62
Transient Ischemic Attack (TIA) (Vascular disorders) | 25
Cerebrovascular Accident (CVA) (Vascular disorders) | 51
Deep Vein Thrombosis (DVT) (Vascular disorders) | 12
Pulmonary Embolism (PE) (Vascular disorders) | 16
Distal thromboemboli (Vascular disorders) | 1
Pericardial effusion - unrelated procedure/device (Cardiac disorders) | 3
Pericarditis - unrelated procedure/device (Cardiac disorders) | 4
Hematoma - unrelated procedure/device (Vascular disorders) | 3
Hemorrhage - unrelated procedure/device (Vascular disorders) | 1
Patient Condition - Non-Cardiovascular - OTHER (General disorders) | 47
Death (General disorders) | 38
System Infection (Infections and infestations) | 76
Fever and/or Virus (Infections and infestations) | 6
Physical Trauma (General disorders) | 76
Abnormal Laboratory Values (General disorders) | 36
Hematological (Blood and lymphatic system disorders) | 39
Neurological (Nervous system disorders) | 54
Gastrointestinal (Gastrointestinal disorders) | 188
Pulmonary (Respiratory, thoracic and mediastinal disorders) | 183
Genitourinary (Renal and urinary disorders) | 50
Renal (Renal and urinary disorders) | 108
Musculoskeletal (Musculoskeletal and connective tissue disorders) | 83
Psychological (Psychiatric disorders) | 8
Integumentary (Skin and subcutaneous tissue disorders) | 39
Head, eyes, ears, nose, throat (HEENT) (General disorders) | 37
Endocrine (Endocrine disorders) | 27
Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 68
Multi-System Failure (General disorders) | 8
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | RELIANCE 4-SITE (N=1820)
Oversensing - RA (Product Issues) | 8
Unable to Capture - RA (Product Issues) | 1
Other - PG System (Product Issues) | 1
Oversensing - RV 1120 - Undersensing - RV (Product Issues) | 2
Elevated Threshold - RV (Product Issues) | 4
Elevated Threshold - LV (Product Issues) | 3
Extracardiac Stimulation - LV (Product Issues) | 7
Inappropriate Tachy Therapy - SVT (Product Issues) | 43
Inappropriate Tachy Therapy - Other (Product Issues) | 11
Early ERI - Premature declaration (Product Issues) | 1
Pacemaker Mediated Tachycardia (PMT) (Product Issues) | 6
Infection (> 30 days post implant) (Infections and infestations) | 3
Psychological effect due to device therapy (Psychiatric disorders) | 3
Hematoma- Pocket (>30 days post implant) (Injury, poisoning and procedural complications) | 1
Seroma - Pocket (>30 days post implant) (Injury, poisoning and procedural complications) | 1
Migration (Injury, poisoning and procedural complications) | 3
Post Surgical wound discomfort/bruising/swelling (Injury, poisoning and procedural complications) | 82
Post-surgical pocket hemorrhage/bleeding/drainage (Injury, poisoning and procedural complications) | 4
Post -Surgical infection (≤ 30 days post implant) (Injury, poisoning and procedural complications) | 6
Adverse Reaction - General (Injury, poisoning and procedural complications) | 10
Adverse Reaction - Respiratory (Injury, poisoning and procedural complications) | 2
Adverse Reaction - Bradycardia (Injury, poisoning and procedural complications) | 1
Adverse Reaction - Hypotension (Injury, poisoning and procedural complications) | 3
Inadvertent VT/VF (Injury, poisoning and procedural complications) | 1
Chest pain (Injury, poisoning and procedural complications) | 6
Physical trauma (Injury, poisoning and procedural complications) | 5
Hematoma - pocket (≤ 30 days post-implant) (Injury, poisoning and procedural complications) | 72
Seroma - Pocket (≤ 30 days post implant) (Injury, poisoning and procedural complications) | 2
Thromboembolic events (Injury, poisoning and procedural complications) | 9
Procedure - PG System - Other (Injury, poisoning and procedural complications) | 9
Oversensing - RA (Product Issues) | 3
Undersensing - RA 2032 - Unable to Capture - RA (Product Issues) | 1
Elevated Threshold - RA (Product Issues) | 2
Extracardiac Stimulation - RA (Product Issues) | 2
Conductor Coil Fracture - RA (Product Issues) | 1
High Out of Range Impedance - RA (Product Issues) | 1
Dislodgement - Multiple signs- RA (Product Issues) | 1
Dislodgement - No reported signs - RA (Product Issues) | 4
Other Lead Related (Product Issues) | 7
Oversensing - RV (Product Issues) | 7
Undersensing - RV (Product Issues) | 2
Unable to Capture - RV (Product Issues) | 1
Elevated Threshold - RV 2140 - Extracardiac Stimulation - RV (Product Issues) | 12
Extracardiac Stimulation - RV (Product Issues) | 4
Myocardial Perforation post implant- RV (Product Issues) | 2
Low Out of Range Impedance - RV (Product Issues) | 2
Dislodgement - Unable to capture - RV (Product Issues) | 3
Dislodgement - Elevated threshold - RV (Product Issues) | 3
Dislodgement - Oversensing- RV (Product Issues) | 1
Dislodgement - Multiple signs - RV (Product Issues) | 2
Dislodgement - No reported signs - RV (Product Issues) | 3
Unable to Capture - LV (Product Issues) | 3
Elevated Threshold - LV (Product Issues) | 8
Extracardiac Stimulation - LV (Product Issues) | 29
Low Out of Range Impedance - LV (Product Issues) | 1
Dislodgement - Unable to Capture - LV (Product Issues) | 1
Dislodgement - No reported signs - LV (Product Issues) | 1
Unable to Convert (Product Issues) | 1
Inappropriate tachy therapy - SVT (Product Issues) | 1
Inappropriate tachy therapy - Noise (Product Issues) | 1
Puncture Site hematoma (Injury, poisoning and procedural complications) | 1
Pneumothorax (Injury, poisoning and procedural complications) | 2
Pleural effusion (Injury, poisoning and procedural complications) | 1
Sinus Bradycardia (Cardiac disorders) | 2
Chronotropic Incompetence (Cardiac disorders) | 1
Ventricular Fibrillation (VF) (Cardiac disorders) | 24
Ventricular Tachycardia (VT)/Monomorphic VT (Cardiac disorders) | 73
Torsades de Pointes (Cardiac disorders) | 1
Nonsustained ventricular tachycardia (NSVT) (Cardiac disorders) | 54
Atrial Fibrillation (AF) (Cardiac disorders) | 111
Atrial Flutter (Cardiac disorders) | 28
Sinus Tachycardia (Cardiac disorders) | 4
Atrial Tachycardia/Other SVT (e.g. AVRT, AVNRT, EAT) (Cardiac disorders) | 25
Premature Ventricular Contractions (PVC) (Cardiac disorders) | 17
Syncope - Heart Failure (Cardiac disorders) | 1
Dizziness - Heart Failure (Cardiac disorders) | 1
Chest Pain - Heart Failure (Cardiac disorders) | 4
Dyspnea - Heart Failure (Cardiac disorders) | 49
Peripheral edema - Heart Failure (Cardiac disorders) | 39
Pulmonary Edema - Heart Failure (Cardiac disorders) | 4
Fatigue - Heart Failure (Cardiac disorders) | 4
Renal Failure/Insufficiency - Heart Failure (Cardiac disorders) | 1
Gastrointestinal - Heart Failure (Cardiac disorders) | 1
Hypotension - Heart Failure (Cardiac disorders) | 1
Weight Gain - Heart Failure (Cardiac disorders) | 6
Heart Failure Symptoms - Unspecified (Cardiac disorders) | 37
Multiple Heart Failure Symptoms (Cardiac disorders) | 75
Hypertension - Heart Failure (Cardiac disorders) | 1
Heart Failure Patient Condition - Cardiovascular - OTHER (Cardiac disorders) | 3
Hypotension/Orthostatic Hypotension (Vascular disorders) | 65
Hypertension/Hypertensive Crisis (Vascular disorders) | 42
Myocardial Infarction (Vascular disorders) | 7
Peripheral Vascular Disease (Vascular disorders) | 27
Intermittent Claudication (Vascular disorders) | 2
Aortic Stenosis (Cardiac disorders) | 1
Aortic Regurgitation (Cardiac disorders) | 2
Mitral Regurgitation (Cardiac disorders) | 6
Syncope (General disorders) | 23
Dizziness (General disorders) | 65
Chest Pain - Ischemic (Vascular disorders) | 14
Chest Pain - Other (General disorders) | 83
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 41
Palpitations (Cardiac disorders) | 16
Fatigue/Weakness (General disorders) | 39
Patient Condition - Cardiovascular - OTHER (Cardiac disorders) | 32
Transient Ischemic Attack (TIA) (Vascular disorders) | 5
Cerebrovascular Accident (CVA) (Vascular disorders) | 3
Deep Vein Thrombosis (DVT) (Vascular disorders) | 12
Pulmonary Embolism (PE) (Vascular disorders) | 1
Distal thromboemboli (Vascular disorders) | 2
Intracardiac thrombus (Cardiac disorders) | 8
Pericardial effusion - unrelated procedure/device (Cardiac disorders) | 1
Pericarditis - unrelated procedure/device (Cardiac disorders) | 2
Hematoma - unrelated procedure/device (Vascular disorders) | 6
Patient Condition - Non-Cardiovascular - OTHER (General disorders) | 109
System Infection (Infections and infestations) | 7
Fever and/or Virus (Infections and infestations) | 1
Physical Trauma (General disorders) | 97
Abnormal Laboratory Values (General disorders) | 95
Hematological (Blood and lymphatic system disorders) | 34
Neurological (Nervous system disorders) | 67
Gastrointestinal (Gastrointestinal disorders) | 166
Pulmonary (Respiratory, thoracic and mediastinal disorders) | 123
Genitourinary (Renal and urinary disorders) | 95
Renal (Renal and urinary disorders) | 74
Musculoskeletal (Musculoskeletal and connective tissue disorders) | 165
Psychological (Psychiatric disorders) | 29
Integumentary (Skin and subcutaneous tissue disorders) | 99
Head, eyes, ears, nose, throat (HEENT) (General disorders) | 185
Endocrine (Endocrine disorders) | 58
Immune (Immune system disorders) | 7
Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 34

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2012-11-02): https://cdn.clinicaltrials.gov/large-docs/95/NCT01596595/Prot_SAP_000.pdf